CLINICAL TRIAL: NCT01965067
Title: A Randomized, Parallel-group, Safety-assessor-blinded Phase IV Study to Estimate the Influence of Mild Hypothermia on Reversal of Rocuronium-induced Neuromuscular Block With Sugammadex
Brief Title: Influence of Mild Hypothermia on Reversal of Rocuronium With Sugammadex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MSD Korea Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MK8616-099
Record Dates: First submitted 2013-10-09; First posted 2013-10-18 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-07

CONDITIONS: Underdosing of Other General Anesthetics
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- C group (Active Comparator): normal thermal condition with core temperatures between 36.5°C and 37°C
  Interventions: Drug: sugammadex
- H group (Experimental): mild hypothermia with core temperatures between 34.5°C and 35°C
  Interventions: Drug: sugammadex

INTERVENTIONS:
Drug: sugammadex — sugammadex 4.0 mg/kg is administered in deep block state(1 - 2 PTCs) in different temperature state
  Reversal effect of sugammadex in temperature state

SUMMARY:
The primary efficacy endpoint is the time from the start of administration of sugammadex to recovery of the TOF ratio to 0.9 in deep neuromuscular block (1-2 twitches post-tetanic count) induced by rocuronium during mild hypothermia with core temperatures between 34.5°C and 35°C, and compared with the normal thermal condition.

Secondary endpoints include time from the start of administration of sugammadex to recovery of the TOF ratio to 0.7 or 0.8 in both groups, vital signs [heart rate and blood pressure] at pre-reversal, post-reversal, recovery and post-anesthetic visit, the incidence of residual neuromuscular blockade, post-operative nausea and vomiting (PONV) and adverse events during mild hypothermia and the normal thermal condition.

We hypothesize that mild hypothermia with core temperatures between 34.5°C and 35°C diminish the efficacy of sugammadex.

DETAILED DESCRIPTION:
This randomized, parallel-group, safety-assessor-blinded phase IV study will be conducted. The study is conducted in accordance with principles of Good Clinical Practice and is approved by the appropriate Institutional Review Boards and regulatory agencies. Written informed consent is obtained from all patients.

In total, 60 patients, aged from 20 to 65 years, with an American Society of Anesthesiologists physical status of I or II and undergoing elective abdominal surgery with a general anesthesia in the supine position will be studied. Patients are excluded if they are expected to have a difficult airway, known neuromuscular disease, significant hepatic or renal dysfunction, family history of malignant hyperthermia, known allergy to one of the drugs used in this protocol, intake of any medication that might interact with muscle relaxants, pregnant, or breast feeding.

The anesthetized patients are randomly assigned to 2 groups as normal thermal condition with core temperatures between 36.5°C and 37°C (C group) and mild hypothermia with core temperatures between 34.5°C and 35°C (H group) in deep block state (1-2 twitches post-tetanic count). The randomization is performed by using computer-generated sealed envelopes to determine which condition (normal thermal condition or mild hypothermia) the patients are performed during deep block state (1-2 twitches post-tetanic count). The anesthesiologist remains blinded to the C group or H group during deep block state (1-2 twitches post-tetanic count) given throughout the remaining course of anesthesia. No premedication is given. After arrival to the operating room, electrocardiography, non-invasive measurement of blood pressure and oxygen saturation are performed. All patients are connected to a bispectral index (BIS) monitor (Model A 2000, Aspect Medical Systems, Natick, MA, USA). Anesthesia is induced with remifentanil 0.5 μg/kg/min injected intravenously over 120 seconds (s) followed by propofol 2 - 2.5 mg/kg injected intravenously over 30 s. After loss of consciousness and ventilation via facemask with a fresh gas flow at 4 L/min (50% nitrous oxide in oxygen) control manually to maintain the end-tidal carbon dioxide (CO2) at 30 to 35 mmHg. Maintenance of anesthesia is with 1 - 1.5 minimum alveolar concentration (MAC) of sevoflurane in a gas mixture of 50% nitrous oxide in oxygen to maintain a BIS between 40 and 50 and infusion doses of remifentanil 0.05 - 0.2 μg/kg/min throughout surgery.

Core body temperature is measured by a thermocouple placed in the distal esophagus (DeRoyal®, DeRoyal Industries Inc., Powell, TN, USA). Core temperature is manipulated in core temperature ranges: 36.5°C and 37°C in C group and 34.5°C and 35°C in H group by surface cooling with wet towels and a fan of air conditioner. The target temperature, once achieved and stabilized, is maintained within ± 0.1°C throughout the remainder of the study. The peripheral skin temperature on the wrist is maintained more than 32°C in both groups.

Neuromuscular function is assessed using acceleromyography of the adductor pollicis muscle (TOF-Watch SX®, Organon Ltd., Dublin, Ireland). Before placing the surface electrodes, the skin overlying the ulnar nerve of the dominant hands is cleansed with isopropyl alcohol. Two electrodes (CleartrodeTM, Ref 1720-003, ConMed®, Utica, NY, USA) are placed over the prepared skin on the wrist. A force displacement transducer is attached to the thumb. No special arm board is used and no preload is applied to the thumb during the entire study procedure.

After the loss of eyelash reflex is confirmed, neuromuscular monitoring begins immediately. For the calibration of acceleromyography, a 5-s 50-Hz supramaximal tetanic stimulus is administered over the ulnar nerve. Calibration is done using the CAL2 mode of the TOF-Watch SX. A supramaximal current is obtained after the initial single twitch calibration. After stabilization of control responses, rocuronium (0.6 mg/kg) is administered and tracheal intubation is performed at the disappearance of the TOF response. Ventilation is adjusted to maintain end-tidal carbon dioxide between 30 and 35 mm Hg. Train-of-four (TOF) stimulation (0.2 ms duration, frequency 2 Hz, 2 s duration with supramaximal current) is performed every 15 s. When no TOF response could be detected, the investigators performed post-tetanic count (PTC) stimulation manually every 6 min to monitor more profound neuromuscular block. As soon as muscle relaxation is no longer required after surgical dressing and the TOF-Watch SX reading is 1 - 2 PTCs, a single IV bolus dose of sugammadex 4.0 mg/kg is administered in deep block state. After the recovery of the TOF ratio to 0.9 is completely confirmed, inhalation agent is finished. Extubation is carried out after confirming the recovery of consciousness and regular respiration. All neuromuscular data are collected on a computer and monitored throughout the study. Skin temperature on the wrist is maintained to more than 32°C using a wrapping cotton wool.

Each patient is monitored for safety for up to 7 days after administration of the study drug. Safety variables comprise all reported adverse events (AEs)(including serious AEs), coded using the Medical Dictionary for Regulatory Activities, vital signs, physical examination, and clinical evidence of residual neuromuscular block (NMB) and recurrence of NMB. A blinded safety assessor performs the safety assessments in the post-operative period and in the follow-up period. The anesthesiologist administering the anesthesia during the surgical procedure is not blinded to the randomized study drug, but the safety assessor is not allowed to reveal the assigned treatment group.

Risk factors for post-operative nausea and vomiting (PONV) are also assessed at baseline and used to assess the likelihood that any occurrences of PONV are associated with study therapy. Subsequent incidence of PONV is determined from AEs coded with the Medical Dictionary for Regulatory Activities preferred terms of nausea, procedural nausea, vomiting and procedural vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Patient for elective abdominal surgery from 20 years (yrs) to 65 yrs Patient in American Society of Anesthesiologists criteria 1 or 2 Patient in the supine position with arm available for neuromuscular monitoring during operation

Exclusion Criteria:

* Patients expected to have a difficult airway, known neuromuscular disease, significant hepatic or renal dysfunction, family history of malignant hyperthermia, known allergy to one of the drugs used in this protocol, intake of any medication that might interact with muscle relaxants, pregnant, or breast feeding

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyo Sang Kim, MD, PhD, Principal Investigator — Department of Anesthesiology and Pain Medicine, Hanyang University Hospital
Locations (1):
- Department of Anesthesiology and Pain Medicine, Hanyang University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee HJ, Kim KS, Jeong JS, Kim KN, Lee BC. The influence of mild hypothermia on reversal of rocuronium-induced deep neuromuscular block with sugammadex. BMC Anesthesiol. 2015 Jan 21;15:7. doi: 10.1186/1471-2253-15-7. PMID 25971394

RESULTS

PARTICIPANT FLOW:
Groups:
- C Group: normal thermal condition with core temperatures between 36.5°C and 37°C
  sugammadex: sugammadex 4.0 mg/kg is administered in deep block state(1 - 2 PTCs) in different temperature state
  Reversal effect of sugammadex in temperature state
- H Group: mild hypothermia with core temperatures between 34.5°C and 35°C
  sugammadex: sugammadex 4.0 mg/kg is administered in deep block state(1 - 2 PTCs) in different temperature state
  Reversal effect of sugammadex in temperature state
Period: Overall Study
Arm/Group | C Group | H Group
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | H Group | C Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (9.8) | 47.4 (9.4) | 47.5 (9.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Reversal Time of Rocuronium
Description: The time from the administration of sugammadex to recovery of the TOF ratio to 0.9 in deep neuromuscular block (1-2 twitches post-tetanic count) induced by rocuronium during mild hypothermia with core temperatures between 34.5°C and 35°C, and compared with the normal thermal condition.
Time Frame: The recovery time to the TOF ratio of 0.9 after the administration of the sugammadex, an expected average of 5 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | C Group | H Group
Number analyzed (Participants) | 30 | 30
seconds | 124.9 (59.2) | 171.1 (62.1)

2. Other Pre Specified Outcome: Incidence of Residual Neuromuscular Blockade
Time Frame: During 1day after operation
Measure: Number; unit: participants
Arm/Group | C Group | H Group
Number analyzed (Participants) | 30 | 30
participants | 0 | 0

3. Other Pre Specified Outcome: Post-operative Nausea and Vomiting
Time Frame: During 7days after operation
Measure: Number; unit: participants
Arm/Group | C Group | H Group
Number analyzed (Participants) | 30 | 30
participants | 0 | 0

4. Other Pre Specified Outcome: Adverse Events
Description: adverse effect of sugammadex(hypersensitivity, dry mouth, hypertension etc.)
Time Frame: During 7days after operation
Measure: Number; unit: participants
Arm/Group | C Group | H Group
Number analyzed (Participants) | 30 | 30
participants | 0 | 0

5. Secondary Outcome: Mean Arterial Blood Pressure
Description: From the start of administration of sugammadex to recovery of the TOF ratio to 0.7 or 0.8 in both groups, mean arterial blood pressure at 1 min before reversal(pre-reversal), 1 min after reversal(post-reversal), recovery and 1 day after surgery (post-anesthetic visit).
Time Frame: 1 min before reversal, 1 min after reversal, 1 day after surgery
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | C Group | H Group
Number analyzed (Participants) | 30 | 30
mmHg
  Mean arterial pressure at 1 min before reversal | 89.9 (10.6) | 91.6 (9.1)
  Mean arterial pressure at 1 min after reversal | 88.4 (10.5) | 89.6 (10.1)
  Mean arterial pressure at 3 min after reversal | 87.5 (11.5) | 90.2 (13.7)
  Mean arterial pressure at 1 day after surgery | 95.0 (12.4) | 94.6 (8.5)

6. Secondary Outcome: Heart Rate
Description: From the start of administration of sugammadex to recovery of the TOF ratio to 0.7 or 0.8 in both groups, Heart rate at 1 min before reversal(pre-reversal), 1 min after reversal(post-reversal), recovery and 1 day after surgery (post-anesthetic visit).
Time Frame: 1 min before reversal, 1 min after reversal, 1 day after surgery
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | C Group | H Group
Number analyzed (Participants) | 30 | 30
beats/min
  Heart rate at 1 min before reversal | 77.5 (10.4) | 77.8 (8.7)
  Heart rate at 1 min after reversal | 71.8 (10) | 72.9 (9.1)
  Heart rate at 3 min after reversal | 70.7 (10) | 73.1 (9.1)
  Heart rate at 1 day after reversal | 81.6 (13.9) | 84.2 (14.8)

ADVERSE EVENTS:
Arm/Group | C Group | H Group
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No